CLINICAL TRIAL: NCT03593928
Title: Pre-intervention and Post-intervention Optical Coherence Tomography Examination for Culprit Lesion in Patients With ST-segment Elevation Myocardial Infarction
Brief Title: Optical Coherence Tomography Examination in Acute Myocardial Infarction
Acronym: OCTAMI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Principal Investigator, hongbing_yan, Co-Director, center of coronary artery disease, Fuwai hospital, China National Center for Cardiovascular Diseases
Other Study IDs: 2018-0710
Record Dates: First submitted 2018-07-11; First posted 2018-07-20 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Myocardial Infarction; Optical Coherence Tomography
Keywords: biomarker; plaque morphology
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma; serum; monocyte
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Different plaque morphology may have an important effect on the prognosis of acute myocardial infarction (AMI), as recent studies show that patients with plaque rupture have a significantly higher risk of cardiac events compared with those with plaque erosion. The primary purpose of this study is to find risk factors and biomarkers for different culprit lesion morphology to perform accurate risk stratification and determine an appropriate treatment strategy for patients with AMI.

DETAILED DESCRIPTION:
Acute myocardial infarction (AMI), which results from coronary artery occlusion due to thrombosis, remains the leading cause of death and disability worldwide. Pathological studies have demonstrated that plaque rupture accompanied by subsequent thrombus formation is the main mechanism responsible for AMI, accounting for approximately two thirds of cases; the remaining approximately one third of cases are the result of plaque erosion. Moreover, previous studies showed that the risk of cardiovascular events is significantly higher in patients with plaque rupture compared to those with plaque erosion. The EROSION study suggested that in patients with acute coronary syndrome presenting with plaque erosion, conservative treatment with anti-thrombotic therapy may be a reasonable option instead of stents implantation. Therefore, it is important to differentiate between the culprit morphologies in order to perform an accurate risk stratification and determine a personalized treatment strategy with the goal to improve the prognosis of patients with AMI.

Optical coherence tomography (OCT), a newly developed high resolution near infrared light-based intravascular imaging modality, can visualize the microstructure of atherosclerotic plaques such as the fibrotic cap, lipid pool, thrombi, and so on, and has been considered as the golden standard for differentiating plaque morphology in vivo.

In this study, we aimed to find risk factors and biomarkers for culprit lesion morphology as assessed by OCT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ST-segment elevation myocardial infarction (defined as continuous chest pain lasted >30 min, ST-segment elevation >0.1 mV in at least two contiguous leads or new left bundle-branch block on the 18-lead electrocardiogram (ECG), and an elevated troponin I level)
* Age ≥18 years
* Provide written informed consent

Exclusion Criteria:

* Cardiac shock
* History of coronary artery bypass graft
* Left main diseases, extremely tortuous or heavily calcified vessels, or chronic total occlusion
* Inability to obtain Thrombolysis in myocardial infarction flow grade ≥ 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (age ≥18 years) who presented with STEMI and underwent emergent procedures were prospectively screened for OCT examination of the culprit lesion.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2017-03-29 (Actual); Primary Completion 2020-03-29 (Estimated); Study Completion 2020-04-29 (Estimated)

PRIMARY OUTCOMES:
culprit lesion morphology as assessed by OCT | 1 day (pre-intervention OCT examination of culprit lesion)
  plaque rupture, plaque erosion or calcified nodule

CONTACTS AND LOCATIONS:
Overall Officials: Hongbing Yan, MD, Principal Investigator — Fuwai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences
Locations (1):
- Chinese Academy of Medical Sciences, Fuwai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li J, Chen R, Zhou J, Wang Y, Zhao X, Liu C, Zhou P, Chen Y, Song L, Yan S, Yan H, Zhao H. Associations of Culprit Vessel Size and Plaque Characteristics in Patients with ST-Segment Elevation Myocardial Infarction. Rev Cardiovasc Med. 2023 Jun 29;24(7):186. doi: 10.31083/j.rcm2407186. eCollection 2023 Jul. PMID 39077009
- [Derived] Zhao X, Zhao H, Chen R, Li J, Zhou J, Li N, Yan S, Liu C, Zhou P, Chen Y, Song L, Yan H. A Combined Measure of the Triglyceride Glucose Index and Trimethylamine N-Oxide in Risk Stratification of ST-Segment Elevation Myocardial Infarction Patients with High-Risk Plaque Features Defined by Optical Coherence Tomography: A Substudy of the OCTAMI Registry Study. Vasc Health Risk Manag. 2024 Mar 29;20:141-155. doi: 10.2147/VHRM.S443742. eCollection 2024. PMID 38567028
- [Derived] Li N, Zhou J, Chen R, Zhao X, Li J, Zhou P, Liu C, Chen Y, Wang Y, Song L, Yan S, Zhao H, Yan H. Prognostic impacts of diabetes status and lipoprotein(a) levels in patients with ST-segment elevation myocardial infarction: a prospective cohort study. Cardiovasc Diabetol. 2023 Jun 26;22(1):151. doi: 10.1186/s12933-023-01881-w. PMID 37365608
- [Derived] Li N, Chen R, Li J, Zhao X, Wang Y, Zhou J, Zhou P, Liu C, Chen Y, Song L, Yan S, Zhao H, Yan H. Prognostic significance of serial N-terminal pro-B-type natriuretic peptide levels in patients with acute myocardial infarction: A prospective study. Am Heart J. 2023 Aug;262:90-99. doi: 10.1016/j.ahj.2023.04.015. Epub 2023 Apr 26. PMID 37116605
- [Derived] Zhao X, Wang Y, Chen R, Li J, Zhou J, Liu C, Zhou P, Sheng Z, Chen Y, Song L, Zhao H, Yan H. Prognostic value of characteristics of plaque combined with residual syntax score among patients with STEMI undergoing primary PCI: an intravascular optical coherence tomography study. Thromb J. 2021 Nov 12;19(1):85. doi: 10.1186/s12959-021-00329-z. PMID 34772417
- [Derived] Wang Y, Zhao X, Zhou P, Liu C, Sheng Z, Li J, Zhou J, Chen R, Chen Y, Song L, Zhao H, Yan H. Plasma Pentraxin-3 Combined with Plaque Characteristics Predict Cardiovascular Risk in ST-Segment Elevated Myocardial Infarction: An Optical Coherence Tomography Study. J Inflamm Res. 2021 Sep 2;14:4409-4419. doi: 10.2147/JIR.S330600. eCollection 2021. PMID 34511975
- [Derived] Wang Y, Zhao X, Zhou P, Liu C, Sheng Z, Li J, Zhou J, Chen R, Chen Y, Song L, Zhao H, Yan H. Residual SYNTAX Score in Relation to Coronary Culprit Plaque Characteristics and Cardiovascular Risk in ST Segment Elevation Myocardial Infarction: an Intravascular Optical Coherence Tomography Study. J Cardiovasc Transl Res. 2022 Feb;15(1):75-83. doi: 10.1007/s12265-021-10152-6. Epub 2021 Jul 9. PMID 34244969
- [Derived] Zhou J, Chen R, Liu C, Zhou P, Li J, Wang Y, Zhao X, Zhao H, Song L, Yan H. Associations of NETs with inflammatory risk and atherosclerotic severity in ST-segment elevation myocardial infarction. Thromb Res. 2021 Jul;203:5-11. doi: 10.1016/j.thromres.2021.04.015. Epub 2021 Apr 19. PMID 33894474
- [Derived] Li J, Tan Y, Zhou P, Liu C, Zhao H, Song L, Zhou J, Chen R, Wang Y, Zhao X, Chen Y, Yan H. Association of Trimethylamine N-Oxide Levels and Calcification in Culprit Lesion Segments in Patients With ST-Segment-Elevation Myocardial Infarction Evaluated by Optical Coherence Tomography. Front Cardiovasc Med. 2021 Feb 24;8:628471. doi: 10.3389/fcvm.2021.628471. eCollection 2021. PMID 33718451
- [Derived] Zhou J, Yu S, Tan Y, Zhou P, Liu C, Sheng Z, Li J, Chen R, Zhao S, Yan H. Trimethylamine N-Oxide Was Not Associated With 30-Day Left Ventricular Systolic Dysfunction in Patients With a First Anterior ST-Segment Elevation Myocardial Infarction After Primary Revascularization: A Sub-analysis From an Optical Coherence Tomography Registry. Front Cardiovasc Med. 2020 Dec 23;7:613684. doi: 10.3389/fcvm.2020.613684. eCollection 2020. PMID 33426008
- [Derived] Zhou J, Sheng Z, Liu C, Zhou P, Li J, Chen R, Song L, Zhao H, Yan H. Association between Admission Hyperglycemia and Culprit Lesion Characteristics in Nondiabetic Patients with Acute Myocardial Infarction: An Intravascular Optical Coherence Tomography Study. J Diabetes Res. 2020 Jun 20;2020:1763567. doi: 10.1155/2020/1763567. eCollection 2020. PMID 32685552
- [Derived] Sheng Z, Zhou P, Liu C, Li J, Chen R, Zhou J, Song L, Zhao H, Yan H. Relationships of coronary culprit-plaque characteristics with duration of diabetes mellitus in acute myocardial infarction: an intravascular optical coherence tomography study. Cardiovasc Diabetol. 2019 Oct 19;18(1):136. doi: 10.1186/s12933-019-0944-8. PMID 31629406
- [Derived] Tan Y, Sheng Z, Zhou P, Liu C, Zhao H, Song L, Li J, Zhou J, Chen Y, Wang L, Qian H, Sun Z, Qiao S, Xu B, Gao R, Yan H. Plasma Trimethylamine N-Oxide as a Novel Biomarker for Plaque Rupture in Patients With ST-Segment-Elevation Myocardial Infarction. Circ Cardiovasc Interv. 2019 Jan;12(1):e007281. doi: 10.1161/CIRCINTERVENTIONS.118.007281. PMID 30599768